CLINICAL TRIAL: NCT01590290
Title: Randomized Controlled Cluster Trial of Resident Pay for Performance and Cardiovascular Outcomes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Schutt, MD, Resident, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16033
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pay for performance (Active Comparator)
  Interventions: Other: financial compensation
- no pay for performance (No Intervention)

INTERVENTIONS:
Other: financial compensation — financial monetary reimbursement
  Arms: pay for performance

SUMMARY:
The purpose of this study is to determine if a pay for performance model in contrast to the traditional "fee for service" model may improve the number of patients discharged being treated in accordance with Joint Commission on Health Care JCAHO (a non-for profit organization that accredits health care organizations) standards and standard of care for management of hyperlipidemia

In this study the investigators will evaluate these two models by training resident physicians (doctors in training) on JCAHO core measures and specific criteria related to accepted standard of care for acute myocardial infarction and heart failure. The physicians will be randomized to a pay for performance or a fee for service model. Then a medical record review will be performed on patient records that received a discharge diagnosis of myocardial infarction or heart failure and were cared for by the physician subjects

ELIGIBILITY:
Inclusion Criteria:

* Physician inclusion: Resident physician on the Acute Cardiology Service, the Coronary Care Unit, or the General Medicine Service at the University of Virginia
* Patient inclusion: discharge diagnosis of heart failure or myocardial infarction.

Exclusion Criteria:

* Residents that are part of the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
compliance with composite pay for performance measure | 1 month
  In patients discharged from the Coronary Care Unit, Acute Coronary Care Service, or General Medical Service with the discharge diagnosis of either heart failure or myocardial infarction, there is no difference in the rate of compliance with the composite score (see below; Heart Failure Score or Myocardial Infarction Score) between physicians reimbursed in a pay for performance scheme and those who receive no additional reimbursement.

SECONDARY OUTCOMES:
heart failure composite score | 1 month
  In patients discharged from the Coronary Care Unit, Acute Coronary Care Service, or General Medical Service with the discharge diagnosis of heart failure there is no difference between rate of compliance with Heart Failure Score between physicians reimbursed in a pay for performance scheme and those who receive no additional reimbursement.
myocardial infarction score | 1 month
  In patients discharged from the Coronary Care Unit, Acute Coronary Care Service, or General Medical Service with the discharge diagnosis of myocardial infarction there is no difference between the rate of compliance with Myocardial Infarction Score between physicians reimbursed in a pay for performance scheme and those who receive no additional reimbursement.
readmission rate | 30 days
  In patients discharged from the Coronary Care Unit, Acute Coronary Care Service, or General Medical Service with the discharge diagnosis heart failure there is no difference between 30-day readmission rate between patients that had an appointment less than 7 days and those that did not.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States